CLINICAL TRIAL: NCT06869928
Title: Implementation of the Pain and Irritability of Unknown Origin (PIUO) Pathway in Community Pediatric Practices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Harold Siden, Clinical Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H24-00078
Record Dates: First submitted 2024-06-28; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pain; Irritability; Neuropathic Pain
Keywords: Pain; Irritability; Pediatrics; Community; Neuropathic Pain; Severe Neurological Disabilities; Implementation Science; Patient Engagement
MeSH Terms: conditions — Pain; Neuralgia; Patient Participation

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a hybrid implementation-effectiveness study using a pre-post, quasi-experimental design. This study adheres to a patient-oriented research framework, integrates principles of equity, diversity, inclusion, and decolonization in the research process, and includes an integrated knowledge mobilization plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PIUO Pathway (Other): The PIUO Pathway targets PIUO in an intentional, focused, timely, sequential order of standardized steps to support best outcomes for children with SNI and families.
  The PIUO Pathway is comprised of 2 steps. Step 1 is for the pediatrician to conduct a thorough history that includes a pain history to identify known and unknown sources of past and current pain, and a physical examination. Step 2 is to carry out a series of screening tests to further explore any potential underlying disease or injury if not apparent based on the Step 1 history and physical examination. The standard screening tests may include urinalysis, ultrasound, gastric pH, and bloodwork. Each child proceeds through the Pain Pathway as long as their pain persists but may not go through all steps if their pain source is identified or pain resolves at any stage. The Steps of the Pain Pathway may be refined by the team based on the results of Phase 1 study analysis, which is underway.
  Interventions: Other: PIUO Pathway

INTERVENTIONS:
Other: PIUO Pathway — see arm description.

SUMMARY:
The Pain and Irritability of Unknown Origin (PIUO) Pathway is a clinical pathway that was developed to evaluate and manage unexplained pain and irritability for children with severe neurological impairments (SNI) who cannot verbally communicate 'where it hurts'. The investigators studied the usefulness of the Pathway with families and expert clinicians in 4 centres across Canada. The aim of this Phase 2 study is to determine whether this tool can transfer from hospital research centres into the community. The Pathway will be used by community pediatricians across British Columbia (BC) when they see patients with PIUO. The investigators want to know how well these pediatricians can follow the Pathway. The goal is to create a systematic, cohesive approach to enhance the clinical care for all children with complex medical needs experiencing PIUO.

DETAILED DESCRIPTION:
BACKGROUND: Many children with brain-based developmental disorders and their families, specifically those with SNI, experience on-going and difficult-to-treat PIUO. However, currently, no consensus exists among healthcare providers about how to best approach PIUO, which likely exacerbates the challenges in faced by parents in taking care of their children with SNI experiencing PIUO. The PIUO Pathway was developed to streamline pain management and care for these children, who are among the most vulnerable seen in any hospital or clinic. To-date, the PIUO Pathway has only been used by expert clinicians in complex care, palliative medicine, and pain medicine, and in tertiary pediatric care settings. Community pediatricians are not yet trained to use this tool, which limits access of such care to the tertiary care level and/or through access to specialist supports. Training front-line clinicians, specifically community pediatricians, to use the PIUO Pathway holds the potential to delivering sustained, effective, and quality community care that can better serve and reach this vulnerable population of Canadian children and families.

AIMS: To advance the assessment and treatment of PIUO in children with SNI and their families, the primary aims and respective research questions of this hybrid implementation-effectiveness study are:

Primary Implementation Aim 1: To determine the feasibility and effectiveness of, and factors that influence implementing the Pain Pathway. Specifically, do the implementation strategies show promise in facilitating the implementation of the Pain Pathway in community practice?

Primary Intervention Aim 2: To assess the effectiveness of the Pain Pathway intervention on relevant outcomes of children with SNI and their families. Specifically, does the Pain Pathway work to help manage PIUO for children with SNI presenting and their families when seen in a community practice?

METHODS

Study Design

The investigators will conduct a hybrid implementation-effectiveness feasibility study using a pre-post, quasi-experimental design. The study will run from 2023 to 2025. Since the Pain Pathway's effectiveness has not been tested previously in a community pediatric practice setting, the investigators selected a Type 2 hybrid effectiveness-implementation design to determine if the Pain Pathway can be feasibly implemented in a real-world (community-based) setting, while further testing the effectiveness of the intervention under a different condition. A hybrid design can offer a more rapid and efficient means to gather information on the effectiveness of the implementation and intervention, as well as to translate knowledge to practice.

Implementation will be guided by the National Implementation Research Network (NIRN)'s Active Implementation Frameworks. The Active Implementation Frameworks (AIF) is an evidence-based set of process frameworks used to facilitate the successful implementation of innovation into practice, including the delivery of evidence-based health services. The investigators will also refer to the NIRN Implementation Stages Planning Tool to support implementation development. Implementation will be conducted in an integrated, non-linear process across the four stages of the AIF: Stage 1 - Exploration; Stage 2 - Installation; Stage 3 - Initial Implementation; and Stage 4 - Full Implementation. Conducting implementation activities in a stepwise manner will allow the investigators to study the implementation in its entirety, including planning, preparing, training, evaluation, and sustainability.

The investigators will use the Theoretical Domains Framework (TDF) to identify barriers and facilitators to implementation. The investigators will also refer to the Behavioural Change Wheel (BCW) to identify priority mechanisms of action that underlie the selection of implementation strategies, which will target the priority barriers and facilitators that the investigators identify.

The Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework will be used to evaluation implementation processes and outcomes. RE-AIM is an integrated framework developed to support the adoption and sustainable implementation of evidence-based interventions in a wide range of health, public health, and community settings.

Intervention Components

The intervention being implemented consists of two components:

1. Pain Pathway: The Pain Pathway targets PIUO in an intentional, focused, timely, sequential order of standardized steps to support best outcomes for children with SNI and families. It is comprised of 2 steps. Step 1 asks the pediatrician to conduct a thorough history that includes a pain history to identify known and unknown sources of past and current pain, and a physical examination. Step 2 involves carrying out a series of screening tests to explore any potential underlying disease or injury, if not apparent based on Step 1. These tests may include urinalysis, ultrasound, gastric pH, and bloodwork. Each child proceeds through the Pain Pathway as long as their pain persists, but may not go through all steps if their pain source is identified or pain resolves at any stage. The steps of the Pain Pathway may be refined by the study team based on the results of Phase 1 study analysis (NCT03464773), which is underway.
2. Nursing Support: An observation made in the pilot and again in the Phase 1 RCT was that the nurse-family interaction that was provided was perceived to be therapeutic both in cases where a treatable pain source was identified, and in cases when they were not. Therefore, elucidating the impact of nursing support and the nurse-family interaction on patient and family outcomes will be an important intervention evaluation component of this study. A central study nurse will be available to work closely with and consult with community pediatricians at each clinic. Nursing support will be defined as any contact or interaction with families in the context of delivering the Pain Pathway, including communication, consultation, psychosocial support, and service and resource coordination, and quality of and satisfaction with nurse-family interaction as reported by parents of children with SNI partaking in the Pain Pathway.

Hypothesized Mechanisms of Change and Implementation Strategies

The implementation strategies will be developed based on the results of the TDF-guided barrier and facilitator assessment of BC community paediatricians. The investigators will select empirically supported implementation strategies to fulfill each mechanism of action identified as relevant through the BCW, while targeting priority barriers and facilitators. The investigators hypothesize that the intervention functions of education, training, and modeling will likely form the foundation of the implementation strategies because the investigators anticipate that barriers to implementation will include a lack of knowledge of the Pain Pathway (knowledge - education) and how to apply it to practice (training), as well as the limited number of pediatricians with expertise in complex care, pediatric pain, and palliative medicine (lack of confidence in managing complex pain - modelling).

ELIGIBILITY:
Pain Pathway Intervention Inclusion Criteria:

* Children aged 6 months to 18 years with SNI (from any cause) with unexplained pain and irritability and whose cognitive or communication impairments prevent determination of pain location, cause, and type will be eligible to participate.
* Eligible children will have cognitive impairment or be non-verbal. Parents should have sufficient English skills, or have access to assistance, to participate in the clinic visits and complete survey tools.

Pain Pathway Intervention Exclusion Criteria:

* Children not within the specified age range
* Children with communication capabilities and cognitive development to localize their pain
* Children that have an explained and treatable cause of pain and irritability. Parents that do not have sufficient English skills, or have access to assistance, to participate in the clinic visits and complete survey tools.

Implementation Participant Inclusion Criteria:

* General pediatricians
* Practicing in a community clinic in British Columbia

Implementation Participant Exclusion Criteria:

- Healthcare professionals who are not general pediatricians (e.g., pediatrician specialists, nurse practitioners, nurses, other allied health professionals)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Implementation Adoption | End of the Pain Pathway, an average of 1 year to 18 months
  Adoption of the Pain Pathway will be measured by completion rates, self-reported by community pediatricians.
Implementation Reach | Baseline and end of the Pain Pathway, an average of 1 year to 18 months
  Reach of the Pain Pathway will be measured by recruitment and retention rates of community pediatricians, self-reported by community pediatricians.
Implementation Acceptability | End of the Pain Pathway, an average of 1 year to 18 months
  Acceptability of the Pain Pathway will be measured by level of satisfaction (e.g., 1 = very unsatisfied; 7 = very satisfied) based on a Likert scale and self-reported by community pediatricians. Scores will be averaged and higher scores reflect higher levels of satisfaction/acceptability.
PIUO Pain Pathway Effectiveness | End of the Pain Pathway, an average of 1 year to 18 months
  Effectiveness of the PIUO Pain Pathway will be measured by proportion of children with SNI and families who received appropriate steps of investigation and treatment options based on following the steps of the PIUO Pain Pathway.

SECONDARY OUTCOMES:
Pain and Irritability (PIUO) | Baseline and end of the Pain Pathway, an average of 1 year to 18 months
  Number of participants whose pain and irritability (PIUO) scores are lower over time, measured by the parent-reported Pain Survey.
Family Well-being | Baseline and end of the Pain Pathway, an average of 1 year to 18 months
  Family well-being, measured by standardized measures of well-being (e.g., PROMIS-57; 1 = unable to do; 5 = without any difficulty) based on parent/caregiver-report of their child and family unit (scoring min. = 8 and max. = 40). Scores are converted to T-scores (mean T-score = 50; standard deviation = 10).
Factors Influencing Implementation | Baseline and end of the Pain Pathway, an average of 1 year to 18 months
  Factors influencing implementation, including barriers and facilitators and health equity-related, will be measured by identification of these factors through survey and interviews with community pediatricians.

CONTACTS AND LOCATIONS:
Overall Officials: Hal Siden, MD, Principal Investigator — University of British Columbia and BC Children's Hospital Research Institute
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No